CLINICAL TRIAL: NCT02339701
Title: A Randomized, Open Label, Phase II Study: Stereotactic Body Radiotherapy (SBRT) vs Conventional Intensity-modulated Radiotherapy (IMRT) for Low or Intermediate Risk Prostate Cancer in Asia Population
Brief Title: Stereotactic Body Radiotherapy vs Intensity-modulated Radiotherapy in Prostate Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Comprehensive Clinical Trial Unit, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PST005
Record Dates: First submitted 2015-01-13; First posted 2015-01-15 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMRT (Other): Patients will receive 38 fractions of radiation, each fraction size will be 2Gy. The total dose will be 78Gy to PTV 1. Whereas the total dose will be 70Gy over 38 fractions to PTV 2. The treatment will be delivered 5 fractions per week consecutively except public holiday, and the total duration of treatment will be 7.5 to 8 weeks.
  Interventions: Radiation: IMRT
- SBRT (Other): Patients will receive 5 fractions of radiation; each fraction size will be 7.25Gy. The total dose will be 36.25 Gy to PTV1. Whereas the total dose will be 32.5Gy over 5 fractions to PTV2. The 5 treatments will be scheduled to be delivered twice aweek over approximately 15-17 days. A minimum of 72 hours and a maximum of 96 hoursshould separate each treatment. No more than 2 fractions will be delivered per week. The total duration of treatment will be no shorter than 15 days and no longer than 17 days.
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: IMRT
  Arms: IMRT
Radiation: SBRT
  Arms: SBRT

SUMMARY:
The primary goal of this phase II study is to compare the change of EPIC HRQOL scores (1-year minus baseline) between SBRT and IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of prostate adenocarcinoma
* Low or intermediate risk prostate cancer patients (i.e. T1-T2c and PSA 20 and Gleason score < 8) with the risk of pelvic node metastasis 15% as calculated by Roach's formula
* ECOG performance score 0-1
* Age ≥ 18
* History/physical examination within 2 weeks prior to registration
* Able to sign informed-consent

Exclusion Criteria:

* Patients with previous diagnosis of cancer other than prostate cancer and non-melanoma skin cancer.
* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or HIFU for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as LHRH agonists (e.g., goserelin, leuprolide) or LHRHantagonists (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g.DES), or surgical castration (orchiectomy)
* Unstable angina and/or congestive heart failure requiring hospitalization, transmural myocardial infarction within the last 6 months, acute bacterial or fungal infection requiring intravenous antibiotics, chronic obstructive pulmonary disease exacerbation or other respiratory illness requiringhospitalization or precluding study therapy at the time of registration
* Patients who have received prior chemotherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2015-01-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
health-related quality of life (HRQOL) | 1 year

SECONDARY OUTCOMES:
the rate of acute and late GI and GU toxicity | 5 years
biochemical-failure free survival | 5 years
disease-specific survival | 5 years
overall survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Poon DMC, Lam D, Wong KCW, Chu CM, Cheung M, Mo F, Suen J, Ng CF, Chan ATC. Prospective Randomized Phase II Study of Stereotactic Body Radiotherapy (SBRT) vs. Conventional Fractionated Radiotherapy (CFRT) for Chinese Patients with Early-Stage Localized Prostate Cancer. Curr Oncol. 2021 Dec 22;29(1):27-37. doi: 10.3390/curroncol29010003. PMID 35049677